CLINICAL TRIAL: NCT01886976
Title: Clinical Study of Chimeric CD(Cluster of Differentiation)138 Antigen Receptor-modified T Cells in Relapsed and/or Chemotherapy Refractory Multiple Myelomas
Brief Title: Treatment of Chemotherapy Refractory Multiple Myeloma by CART-138
Acronym: CART-138
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, principal investigator, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-008
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Immunotherapy, Adoptive; Sensitivity and Specificity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anti-CD138 CAR T cells (Experimental): Patients receive anti-CD138-CAR retroviral vector-transduced autologous or donor-derived T cells on days 0,1, 2 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: CART-138 cells

INTERVENTIONS:
Biological: CART-138 cells
  Other Names: chimeric antigen receptor T cells with specificity for CD138 genetically modified lymphocyte therapy

SUMMARY:
RATIONALE: Placing a tumor antigen chimeric receptor that has been created in the laboratory into patient autologous or donor-derived T cells may make the body build immune response to kill cancer cells.

PURPOSE: This clinical trial is to study genetically engineered lymphocyte therapy in treating patients with CD138 positive multiple myeloma that is relapsed (after stem cell transplantation or intensive chemotherapy) or refractory to further chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and feasibility of the chimeric antigen receptor T cells transduced with the anti-CD138 vector (referred to as CART-138 cells).

II. Determine duration of in vivo survival of CART-138 cells. RT-PCR (reverse transcription polymerase chain reaction) analysis of whole blood and bone marrow will be used to detect and quantify survival of CART-138 TCR zeta:CD137 and TCR (T-cell receptor) zeta cells over time.

SECONDARY OBJECTIVES:

I. For patients with detectable disease, measure anti-myeloma response due to CART-138 cell infusions.

II. To determine if the CD137 transgene is superior to the TCR zeta only transgene as measured by the relative engraftment levels of CART-138 TCR zeta:CD137 and TCR zeta cells over time.

III. Estimate relative trafficking of CART-138 cells in bone marrow.

IV. For patients with stored or accessible myeloma cells, determine myeloma cell killing by CART-138 cells in vitro.

V. Determine if cellular or humoral host immunity develops against the murine anti-CD138, and assess correlation with loss of detectable CART-138 (loss of engraftment).

VI. Determine the relative subsets of CART-138 T cells (Tcm, Tem, and Treg).

OUTLINE: Patients are assigned to 1 group according to order of enrollment.

Patients receive anti-CD138-CAR (coupled with CD137 and CD3 zeta signalling domains)vector-transduced autologous T cells on days 0,1, and 2 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed intensively for 6 months, every 3 months for 2 years, and annually thereafter for 13 years.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with CD138 positive multiple myeloma in patients with no available curative treatment options (such as autologous or allogeneic SCT) who have limited prognosis (several months to < 2 year survival) with currently available therapies will be enrolled.
* CD138 positive multiple myeloma CR can not be achieved after at least 4 prior combination chemotherapy regimens.
* MM in CR(complete remission)2 or CR3 and not eligible for allogeneic SCT because of age, comorbid disease, or lack of available family member or unrelated donor.
* Less than 1 year between last chemotherapy and progression (i.e. most recent progression free interval < 1 year).
* Relapsed after prior autologous or allogenic SCT. MM patients with relapsed or residual disease after at least 1 prior therapy and not eligible for allogeneic SCT.
* Residual disease after primary therapy and not eligible for autologous SCT

  * Expected survival > 12 weeks
  * Creatinine < 2.5 mg/dl
  * ALT(alanine aminotransferase)/AST (aspartate aminotransferase)< 3x normal
  * Bilirubin < 2.0 mg/dl
  * Any relapse after prior SCT will make patient eligible regardless of other prior therapy
  * Adequate venous access for apheresis, and no other contraindications for leukapheresis
  * Voluntary informed consent is given

Exclusion Criteria:

* Pregnant or lactating women
* The safety of this therapy on unborn children is not known. Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion.
* Uncontrolled active infection.
* Active hepatitis B or hepatitis C infection.
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
* Previously treatment with any gene therapy products
* Feasibility assessment during screening demonstrates < 30% transduction of target lymphocytes, or insufficient expansion (< 5-fold) in response to CD3/CD137 costimulation.
* Any uncontrolled active medical disorder that would preclude participation as outlined.
* HIV infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | Until week 24
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment

SECONDARY OUTCOMES:
Anti-myeloma responses to CART-138 cell infusions | up to 24 weeks
  by measuring the changes of aberrant immunoglobulin in serum and multiple myeloma cells in bone marrow.

OTHER OUTCOMES:
in vivo existence of CART-138 | 1 year
  measurement of CART-138 cells in peripheral blood by PCR method

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China